CLINICAL TRIAL: NCT05658796
Title: Telemedicine-delivered Digital Cognitive Behavioral Intervention to Decrease Post-operative Opioid Use Among Patients Undergoing Total Knee or Hip Arthroplasty
Brief Title: RXWell to Decrease Post-Operative Opioid Use in Total Knee or Hip Arthroplasty
Acronym: RxWell
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Pittsburgh (Other)
Collaborators: National Institutes of Health (NIH) (NIH); National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Principal Investigator, Ata Murat Kaynar, Professor, University of Pittsburgh
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: STUDY21120053; R21DA061414-01 (NIH)
Record Dates: First submitted 2022-07-26; First posted 2022-12-21 (Actual); Last update posted 2025-11-05 (Actual); Status verified 2025-08

CONDITIONS: Mood Disorders; Anxiety; Depressive Symptoms; Depression; Anxiety Disorders; Anxiety Depression
MeSH Terms: conditions — Mood Disorders; Anxiety Disorders; Depression

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Control (Active Comparator): No intervention (No RxWell). Subjects will receive standard of care and education regarding potential resources for anxiety and depression. Subjects will complete questionnaires via REDCap assessing primary and secondary outcomes
  Interventions: Behavioral: -RxWell
- Intervention: RxWell (Experimental): RxWell Intervention. Subjects will receive standard of care and digital cognitive behavioral intervention by using the application RxWell. Subjects will complete questionnaires via REDCap assessing primary and secondary outcomes and will complete GAD-7 (Generalized Anxiety Disorder Scale) and PHQ-8 (Patient Health Questionnaire for Depression) every 2 weeks within the RxWell application.
  Interventions: Behavioral: +RxWell
- Control (screen failures) (No Intervention): We will collect data on patient outcomes for patients that did not meet criteria for the RxWell intervention.

INTERVENTIONS:
Behavioral: +RxWell — During the SuRxgWell trial, if a participant is randomized to receive RxWell, they will be provided with an access code that is required to download the app. Once the participant has downloaded the app, they will be paired with a UPMC coach who will guide the person through the sessions using in-app texting to help give them the tools needed to actively cope with anxiety and/or depression. The UPMC coaches are supervised by a licensed UPMC mental health clinician. The participant will have access to the app and coach for six months after they have consented. The digital behavioral tool includes over 30 brief Cognitive Behavioral Therapy (CBT) and mindfulness-based techniques.
  Arms: Intervention: RxWell
Behavioral: -RxWell — Treatment as usual
  Arms: Control

SUMMARY:
It is envisioned that multipronged benefits from this pilot work for the UPMC ISD and its members. It is expected the RxWell platform to provide the following benefits: expansion of the use of RxWell to all UPMC ISD members providing peri-operative mood management with advantage of improved peri-operative outcomes, improving saving for the UPMC ISD by hastening the recovery and decreased resource utilization, and addition to the high-value care of UPMC with this holistic approach to patient perioperative care

DETAILED DESCRIPTION:
The content of the digital behavioral tool was developed based on standard Cognitive Behavioral Therapy (CBT) techniques. An additional layer of support includes a behavioral health coach who provides guidance and motivation throughout the use of the app via in-app text messaging.

This approach has already been tested at UPMC on multiple adult clinical populations. This project represents the first pilot of the digital behavioral tool with perioperative patients

The digital behavioral tool can provide a resource gap by providing preventive mental health services to promote mental health wellness for patients to help reduce the deleterious impact of established mood disorders on recovery following primary total knee replacements including:

* pain and opioid requirement,
* functional recovery,
* decrease complications, and
* reduce resources utilization such as hospital length of stay, postoperative need for visits and the use of rehabilitation.

  1. Determine the feasibility of using RxWell for patients undergoing elective surgery who have mood disorder symptoms using MyUPMC platform and established either at the time of visiting the Center for Perioperative Care (CPC) either in-person or via anesthesia telemedicine services (ATS) in a tertiary care system.
  2. Determine the impact of RxWell-associated improvements in anxiety, depression, and catastrophizing on postoperative outcomes with a special focus on resources utilization.

Subjects who choose to sign electronically will be provided a link via email for REDCap. This link will include an electronic consent document and the ability to sign with a computer cursor, stylus, or their finger depending on the device the subject uses to access this link.

ELIGIBILITY:
Inclusion Criteria for the RXWell Study:

* Adults >18 years
* Scheduled for elective primary total knee arthroplasty (TKA) or hip replacement (THA) at the approved UPMC hospitals
* Moderately high levels of mood disorder symptoms on validated PROMIS measures, defined as a T-score > or = to 60 on PROMIS Anxiety 4a short form and/or PROMIS Depression4a short form

Exclusion Criteria for the RXWell Study:

* Patients undergoing non-elective surgery or secondary arthroplasty
* Active delirium, neurocognitive impairment, or severe intellectual disability
* No access to a smart device (phone or tablet)
* Active alcoholism (defined as daily use of more than 1 liter of wine and /or 3 or more shots of hard liquor) or drug abuse (defined as daily use of illicit drugs)
* Profound mood disorders requiring immediate intervention such as suicidal ideation, defined as a PROMIS Depression score of more than 70
* A PROMIS Anxiety and/or Depression T-score >70, which corresponds to severe anxiety and depression.

  * Patients needing immediate care will be referred to psychiatrists and primary team.

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2023-01-27 (Actual); Primary Completion 2026-12-01 (Estimated); Study Completion 2026-12-30 (Estimated)

PRIMARY OUTCOMES:
Cumulative Opioid Consumption in Oral Morphine Equivalent (OME) (mg) | POD 1 to Week 4 Post-Op
  This outcome will be measured by extracting pain medication data from the electronic health record to determine OME (oral morphine equivalents) (mg) for opioid medications on POD 1 and 2, and weeks 1 and 4 following surgery. This will be recorded for each study arm as mean (SD).

SECONDARY OUTCOMES:
Opioid prescription refills by 3 months | Post-Op Month 3
  This outcome will be measured by abstracting the PDMP review from the medical records to determine the number of opioid prescription refills by post-op month 3. This will be counted per patient and each arm will be recorded as a mean (SD).
Pain at Rest | Post-Op Day 1, Post-Op Day 2, and Post-Op Day 7
  Pain scores will be collected using a numerical rating scale (NRS) in which 0 = no pain at all, and 10 = worst pain imaginable. This outcome will be averaged in each arm and reported as mean (SD) for each timepoint provided in the time frame.
Pain with Movement | Post-Op Day 1, Post-Op Day 2, and Post-Op Day 7
  Pain scores will be collected using a numerical rating scale (NRS) in which 0 = no pain at all, and 10 = worst pain imaginable. This outcome will be averaged in each arm and reported as mean (SD) for each timepoint provided in the time frame.
Persistent Opioid Use | Post-Op 1 Month, Post-Op 3 Months
  This outcome will be measured by the number of participants still using opioids at the timepoints provided in the time frame. This is a binary yes/no response - yes, the subject is using opioids, no the subject is not using opioids and will be abstracted from the medical records.

CONTACTS AND LOCATIONS:
Overall Officials: Ata Murat Kaynar, MD, MPH, Principal Investigator — UPMC Department of Anesthesiology and Perioperative Medicine
Locations (3):
- United States (3):
  - UPMC East, Monroeville, Pennsylvania
  - UPMC Shadyside, Pittsburgh, Pennsylvania
  - UPMC Passavant, Pittsburgh, Pennsylvania

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Kaynar AM, Lin C, Sanchez AG, Lavage DR, Monroe A, Zharichenko N, Strassburger M, Saucier K, Groff YJ, Klatt BA, O'Malley MJ, Szigethy E, Wasan AD, Chelly JE. SuRxgWell: study protocol for a randomized controlled trial of telemedicine-based digital cognitive behavioral intervention for high anxiety and depression among patients undergoing elective hip and knee arthroplasty surgery. Trials. 2023 Nov 9;24(1):715. doi: 10.1186/s13063-023-07634-0. PMID 37946291